CLINICAL TRIAL: NCT04818710
Title: Comparative Study Between Scalpel and Diathermy Skin Incision in Repeated Cesarean Section
Brief Title: Scalpel Versus Diathermy Skin Incision in Repeated CS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mazen Abdel Rasheed, Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: diathermy skin incision
Record Dates: First submitted 2021-03-20; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Benifits of Using Diathermy in Skin Incision
MeSH Terms: interventions — Diathermy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- skin incision with a scalpel (Placebo Comparator): In the scalpel group, the incision was made by the traditional method, with proper homeostasis by applying pressure to skin blood vessels and ligating the subcutaneous bleeding.
  Interventions: Procedure: skin incision with a scalpel
- skin incision with diathermy (Active Comparator): In the diathermy group, the incision made using a small flat blade pen electrode, set on cutting mode and delivering a 120 watt (maximum) sinusoidal current, electrosurgical cutting performed without pressure or mechanical displacement.
  Interventions: Procedure: skin incision with diathermy

INTERVENTIONS:
Procedure: skin incision with a scalpel — A Pfannenstiel skin incision was done through the subcutaneous tissue, rectus sheath and dissected from rectus muscle until peritoneum was visualized.
  group 1 (skin incision with a scalpel)
  Arms: skin incision with a scalpel
Procedure: skin incision with diathermy — A Pfannenstiel skin incision was done through the subcutaneous tissue, rectus sheath and dissected from rectus muscle until peritoneum was visualized.
  group 2 (skin incision with diathermy)
  Arms: skin incision with diathermy

SUMMARY:
This study was performed to compare both methods of skin incisions to determine differences in postoperative pain, hemodynamic changes, incisional time, blood loss during incision, wound healing, and wound complication.

DETAILED DESCRIPTION:
Our study aims to compare the use of diathermy versus scalpel in making skin incision during cesarean section to judge the variations in

1. incision time,
2. incision blood loss,
3. hemodynamic changes,
4. postoperative pain,
5. wound healing
6. wound complications.

ELIGIBILITY:
Inclusion Criteria:

* women with a history of only one previous cesarean section
* age between 18 and 40 years
* gestational age of 38 to 41 weeks
* body mass index less than 30.

Exclusion Criteria:

* any medical disorder that can affect wound healing as diabetes, chronic anemia, chronic skin conditions, history of allergy, or history of an infected surgical wound.
* Women who conducted primary or emergency cesarean deliveries
* cardiac patients on pacemakers
* patients on anticoagulants
* women refusing to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 476 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
incision time | during surgical operation. the difference between starting skin incision till the rectus sheath was visualized
  We compared incisional time by using a digital clock. The incisional time was established as follows: when skin incision was made, the surgeon called out "start the clock". Once the rectus sheath was visualized, the surgeon calls out "stop the clock". The incision time was the difference between "start" and "stop".
incision blood loss | during surgery
  This was calculated by weighing the swabs pre and postoperatively (1mg = 1ml) after complete hemostasis was achieved.
postoperative pain | during the first day after surgery
  We compared those patients clinically for postoperative pain for 24 hours by visual analog scale (VAS) score, a psychometric response scale, and it is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. It is 11 points numeric scale ranges from "0" representing one pain extreme (e.g., no pain) to "10" representing the other pain extreme (e.g., "pain as bad as you can imagine" or "worst pain imaginable"). This score was recorded for each participant at 2,4,6,8,10,12,24 hours postoperatively.

SECONDARY OUTCOMES:
wound healing | during the first week after surgery
  healing by primary versus secondary intention
wound complications | during the first week after surgery
  like seroma, hematoma, ecchymosis, dehiscence (separation of the subcutaneous tissues with skin), and infection

CONTACTS AND LOCATIONS:
Locations (1):
- National Research Centre, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes